CLINICAL TRIAL: NCT03170843
Title: Randomized Controlled Trial to Evaluate the Effectiveness and Efficacy of a Sterile Circular Polyethylene Drape Compared to Conventional Surgical Dressing in Prevention of Surgical Site Infection
Brief Title: Circular pOlyethylene Drape in preVention of Surgical Site infEction: A Randomized Controlled Trial
Acronym: COVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, Hyung Jin Kim, Professor, Saint Vincent's Hospital, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OTracSSI
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: The experimental group will be using the plastic wound retractor, while the control group will use a conventional surgical pad for wound protection.
Who Masked: Participant
Masking Description: Each participant will be under the general anesthesia without knowing which group is assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- O-Trac (Experimental): The experimental group will use the plastic ring wound retractor for wound protection during the surgery.
  Interventions: Device: use of plastic ring wound retractor
- Surgical pad (No Intervention): The control group will use a conventional surgical pad for wound protection during the surgery.

INTERVENTIONS:
Device: use of plastic ring wound retractor — the experimental arm will use the plastic ring wound retractor for wound protection.
  Arms: O-Trac

SUMMARY:
This study is to evaluate the effectiveness of the plastic ring wound retractor to reduce the rate of surgical site infection in patients who undergo open abdomen surgery for gastrointestinal tract.

DETAILED DESCRIPTION:
Participants who are determined to undergo open abdomen surgery will be screening for the eligibility first. If eligible and agreed to participate, each participant will be assigned to either the experimental group or control group based on the electronic randomization. The experimental group will use the plastic ring wound retractor, while the control group will use a conventional surgical pad for wound protection method. Each participant will be blind to the randomization result because he/she will be under general anesthesia. Once the surgery is finished, the patient will be assessed on the surgical wound at postoperative day 1, 7, 14, 30. Two groups will be compared for the surgical wound infection rate.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years or less than 75 years
* either elective or emergent surgery for upper GI, small intestine, or colorectal disease
* open laparotomy
* the patient who agrees to participate in this trial

Exclusion Criteria:

* concurrent abdominal wall infection
* open conversion from laparoscopy
* poor nutritional status, NRS 2002 score 3
* combined hepatobiliary operation
* pregnant or breast-feeding state
* severe immunosuppression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
The rate of surgical wound infection | within 30 days postoperative
  The rate of surgical wound infection will be monitored for each group.

CONTACTS AND LOCATIONS:
Overall Officials: HyungJin Kim, MD, Principal Investigator — Eunpyeong St. Mary's Hospital, The Catholic University of Korea
Locations (13):
- South Korea (13):
  - Chonnam National University Hospital, Gwangju, Chonnam
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwondo
  - National Health Insurance Service Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University of Hospital, Suwon, Gyeonggi-do
  - Ujeongbu St Mary's Hospital, The Catholic University of Korea, Uijeongbu-si, Gyeonggi-do
  - Keimyung University Dongsan Medical Center, Daegu, Gyeongsangbukdo
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Chung-Ang University Hospital, Seoul
  - Eunpyeong St. Mary's hospital, Seoul
  - Yeouido St. Mary's hospital, The Catholic University of Korea, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mihaljevic AL, Michalski CW, Erkan M, Reiser-Erkan C, Jager C, Schuster T, Schuhmacher C, Kleeff J, Friess H. Standard abdominal wound edge protection with surgical dressings vs coverage with a sterile circular polyethylene drape for prevention of surgical site infections (BaFO): study protocol for a randomized controlled trial. Trials. 2012 May 15;13:57. doi: 10.1186/1745-6215-13-57. PMID 22587425
- [Result] Mihaljevic AL, Schirren R, Ozer M, Ottl S, Grun S, Michalski CW, Erkan M, Jager C, Reiser-Erkan C, Kehl V, Schuster T, Roder J, Clauer U, Orlitsch C, Hoffmann TF, Lange R, Harzenetter T, Steiner P, Michalski M, Henkel K, Stadler J, Pistorius GA, Jahn A, Obermaier R, Unger R, Strunk R, Willeke F, Vogelsang H, Halve B, Dietl KH, Hilgenstock H, Meyer A, Kramling HJ, Wagner M, Schoenberg MH, Zeller F, Schmidt J, Friess H, Kleeff J. Multicenter double-blinded randomized controlled trial of standard abdominal wound edge protection with surgical dressings versus coverage with a sterile circular polyethylene drape for prevention of surgical site infections: a CHIR-Net trial (BaFO; NCT01181206). Ann Surg. 2014 Nov;260(5):730-7; discussion 737-9. doi: 10.1097/SLA.0000000000000954. PMID 25379844
- [Result] Pinkney TD, Calvert M, Bartlett DC, Gheorghe A, Redman V, Dowswell G, Hawkins W, Mak T, Youssef H, Richardson C, Hornby S, Magill L, Haslop R, Wilson S, Morton D; West Midlands Research Collaborative; ROSSINI Trial Investigators. Impact of wound edge protection devices on surgical site infection after laparotomy: multicentre randomised controlled trial (ROSSINI Trial). BMJ. 2013 Jul 31;347:f4305. doi: 10.1136/bmj.f4305. PMID 23903454
- [Derived] Yoo N, Mun JY, Kye BH, Kim CW, Lee JI, Park YY, Kang BM, Park BK, Kwak HD, Kang WK, Bae SU, Oh HK, Hong Y, Kim HJ. Plastic Wound Protector vs Surgical Gauze for Surgical Site Infection Reduction in Open GI Surgery: A Randomized Clinical Trial. JAMA Surg. 2024 Jul 1;159(7):737-746. doi: 10.1001/jamasurg.2024.0765. PMID 38656413
- [Derived] Yoo RN, Kim HJ, Lee JI, Kang WK, Kye BH, Kim CW, Bae SU, Nam S, Kang BM. Circular pOlyethylene drape in preVEntion of suRgical site infection (COVER trial): study protocol for a randomised controlled trial. BMJ Open. 2020 Jan 22;10(1):e034687. doi: 10.1136/bmjopen-2019-034687. PMID 31974091